CLINICAL TRIAL: NCT02818803
Title: Efficacy of Standardized-propolis Extract (EPP-AF®) Gel Formulation as Buccal Antiseptic in Elderly People
Brief Title: Efficacy of Standardized-propolis Extract (EPP-AF®) Gel Formulation as Buccal Antiseptic
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Financiadora de Estudos e Projetos (Other)
Responsible Party: Principal Investigator, Erica Negrini Lia, Pos doctoral, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1057529
Record Dates: First submitted 2016-06-21; First posted 2016-06-30 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Candidiasis, Oral; Stomatitis, Denture
Keywords: propolis; therapeutic; miconazole; denture stomatitis
MeSH Terms: conditions — Candidiasis, Oral; Stomatitis, Denture | interventions — Propolis; Miconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propolis (Experimental): Standardized-propolis extract (EPP-AF®) oral gel formulation, 3 times a day, for 14 days
  Interventions: Other: Propolis
- Miconazole (Active Comparator): Miconazole 20mg/g oral gel,3 times a day, for 14 days
  Interventions: Drug: Miconazole

INTERVENTIONS:
Other: Propolis
  Arms: Propolis
Drug: Miconazole
  Other Names: Daktarin oral gel
  Arms: Miconazole

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of propolis on the treatment of oral candidiasis, more specifically denture stomatitis. Half of participants will receive a standardized-propolis (EPP-AF®) gel formulation while the other half will receive miconazole gel, both for oral use.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients with denture stomatitis

Exclusion Criteria:

* Recent use of anti fungals or antibiotics(2 months or less), dementia

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change from Newton Score at 14 days | Day 14
  Clinical assessment of buccal lesions localized at hard palate. The score utilized to measure the intensity of lesions will be Newton classification (I - punctate in the palate; II - extensive smooth reddened appearance; III -extensive reddening with hyperplastic growth) and the outcome will be the reduction of Newton's score comparing day 1 with day 14.

SECONDARY OUTCOMES:
Assessment of gel acceptability | Day 7
  Application of hedonic scale on day 7
Assessment of adverse events | Day 7 and 14
  Questioning about rise of adverse events on days 7 and 14
Anti fungal activity | Day 1 and 14
  Colony forming unit count (CFU/mL) on days 1 and 14

CONTACTS AND LOCATIONS:
Overall Officials: Erica N Lia, PhD, Principal Investigator — Faculdade de Medicina de Ribeirão Preto/USP; Gisela M Pina, DDS, Principal Investigator — Unievangelica Anapolis
Locations (2):
- Brazil (2):
  - Unievangelica Anapolis, Anápolis, Goiás
  - Unidade de Pesquisa Clinica HCRP-USP, Ribeirão Preto, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Freires IA, Queiroz VCPP, Furletti VF, Ikegaki M, de Alencar SM, Duarte MCT, Rosalen PL. Chemical composition and antifungal potential of Brazilian propolis against Candida spp. J Mycol Med. 2016 Jun;26(2):122-132. doi: 10.1016/j.mycmed.2016.01.003. Epub 2016 Feb 23. PMID 26916845
- [Result] Santos VR, Gomes RT, de Mesquita RA, de Moura MD, Franca EC, de Aguiar EG, Naves MD, Abreu JA, Abreu SR. Efficacy of Brazilian propolis gel for the management of denture stomatitis: a pilot study. Phytother Res. 2008 Nov;22(11):1544-7. doi: 10.1002/ptr.2541. PMID 18696746
- [Result] Santos VR, Pimenta FJ, Aguiar MC, do Carmo MA, Naves MD, Mesquita RA. Oral candidiasis treatment with Brazilian ethanol propolis extract. Phytother Res. 2005 Jul;19(7):652-4. doi: 10.1002/ptr.1715. PMID 16161031